CLINICAL TRIAL: NCT00290979
Title: Evaluation of Efficacy and Safety of HMR1964 (Insulin Glulisine) in Subjects With Type 1 Diabetes Mellitus; Insulin Lispro Controlled, Open, Randomized, Parallel Group, Non-inferiority Study, for 28 Weeks
Brief Title: Efficacy and Safety of Insulin Glulisine in Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC6167
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Last update posted 2009-08-26 (Estimated); Status verified 2009-03

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: HMR1964, insulin glulisine, Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — insulin glulisine

INTERVENTIONS:
Drug: insulin glulisine

SUMMARY:
* To evaluate non-inferiority in the efficacy of HMR1964 as compared with Insulin lispro in terms of the change in HbA1C from baseline to endpoint.
* To compare the safety of HMR1964 with insulin lispro.

DETAILED DESCRIPTION:
* To compare HMR1964 with insulin lispro in terms of the change in HbA1C from baseline to week 12 and week 28; consecutive change in HbA1C by every 4 weeks, blood glucose parameters, symptomatic hypoglycemia and insulin doses (rapid-acting, basal and total).
* To collect 6-month safety data of HMR1964.

ELIGIBILITY:
Inclusion Criteria:

* Men or women with type 1 diabetes mellitus, an HbA1C range of >=6.0 - =<11.0%, and on a basal-bolus insulin regimen. They must have had at least 1 year of continuous insulin treatment at the date of informed consent.

Exclusion Criteria:

* Subjects who received an oral hypoglycemic agent other than insulin within 4 weeks prior to informed consent
* Subjects who received oral or intravenous corticosteroid within 4 weeks prior to informed consent
* Subjects who were treated with another investigational product within 12 weeks prior to informed consent
* Subjects with likelihood of requiring concomitant treatment during the study period with drugs not permitted by this study protocol
* Subjects with clinically relevant cardiovascular, hepatic, neurologic, endocrine, active cancer, other serious complication or systemic disease making implementation of the protocol or interpretation of the study results difficult
* Subjects who have undergone pancreatectomy or pancreas/islet cell transplant
* Night shift workers
* Subjects unlikely to comply with the study protocol, e.g., inability to periodic return for follow-up visits, and unlikelihood of completing the study
* Subjects who have previously been treated with HMR1964
* Subjects who are pregnant, breast feeding or wish to become pregnant during the study period
* Female subjects who are possibly pregnant [female subjects of reproductive potential who have serum human chorionic gonadotropin (hCG) level > 0.7 mIU/mL as determined by central laboratory, SRL Medisearch Inc., during screening phase]
* Subjects with diabetic retinopathy who received surgical treatments (laser photocoagulation or vitrectomy) within 24 weeks prior to informed consent, or who are expected to have these surgical treatments during the study period
* Subjects with history of alcohol abuse
* Subjects with hypersensitivity to insulin preparations
* Subjects with impaired hepatic function (SGOT or SGPT ³=<80 IU/L determined by central laboratory, SRL Medisearch Inc., during screening phase) or impaired renal function (serum creatinine =<2.0 mg/dL determined by central laboratory, SRL Medisearch Inc., during screening phase)
* Subjects who are judged by the investigator or subinvestigator as inappropriate as the subjects of this study for any other reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2004-12

PRIMARY OUTCOMES:
Non-inferiority in the efficacy and safety of HMR1964 as compared with Insulin lispro

SECONDARY OUTCOMES:
6-month safety data

CONTACTS AND LOCATIONS:
Overall Officials: Masayoshi KOYAMA, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Tokyo, Japan

REFERENCES:
- [Result] Kawamori R, Kadowaki T, Ishii H, Iwasaki M, Iwamoto Y. Efficacy and safety of insulin glulisine in Japanese patients with type 1 diabetes mellitus. Diabetes Obes Metab. 2009 Sep;11(9):891-9. doi: 10.1111/j.1463-1326.2009.01086.x. Epub 2009 Jul 13. PMID 19614947